CLINICAL TRIAL: NCT07339293
Title: Constipation Insoles
Brief Title: The Effect of Constipation Insoles on the Management of Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Associate Professor Dr., Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Constipation Insoles
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Palliative Care; Constipation
Keywords: constipation; palliative care; reflexology; nursing; comfort
MeSH Terms: conditions — Constipation | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients in the experimental group were instructed to walk with the constipation insole for 20 minutes a day for four weeks, starting from the second week
  Interventions: Behavioral: constipation insole; Behavioral: Walk
- Control Group (Other): Patients in the control group were only instructed to walk for 20 minutes a day for four weeks.
  Interventions: Behavioral: Walk

INTERVENTIONS:
Behavioral: constipation insole — Patients in the experimental group were instructed to walk with the constipation insole for 20 minutes a day for four weeks, starting from the second week
  Arms: Experimental Group
Behavioral: Walk — Patients in the control group were only instructed to walk for 20 minutes a day for four weeks

SUMMARY:
Constipation is a common symptom among patients receiving palliative care and significantly affects their quality of life. Effective management of constipation requires both pharmacological and non-pharmacological approaches. Reflexology has been increasingly used as a complementary method for constipation management; however, factors such as the need for a trained reflexology specialist, time limitations, and financial constraints may limit patients' access to this intervention. To overcome these barriers, a constipation insole based on reflexology principles has been developed, which can be easily used by patients either at home or in clinical settings.

This study was designed as a randomized controlled experimental trial to evaluate the effectiveness of a constipation insole in the management of constipation in patients receiving palliative care. During the first week of the study, no intervention was applied in order to assess participants' baseline bowel habits. Starting from the second week, patients in the experimental group were instructed to walk with the constipation insole for 20 minutes per day for a total of four weeks. Patients in the control group were instructed to walk for 20 minutes per day for the same duration, without using the insole.

At baseline, data were collected using the Patient Identification Form and the General Comfort Scale. Throughout the study period, bowel function and constipation-related outcomes were monitored using standardized measurement tools. The Constipation Assessment Scale was planned to be administered every three days, the Constipation Severity Scale daily, and the Bristol Stool Consistency Scale at each defecation. The General Comfort Scale was planned to be re-administered on the 28th day of the intervention period.

The findings obtained from this study are expected to provide evidence regarding the potential role of constipation insoles as a complementary intervention in constipation management for patients in palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteer to participate in the study and are over 18 years of age,
* Patients without any cognitive, mental, or verbal communication impairments,
* Patients receiving palliative care,
* Patients with constipation,
* Patients with fewer than 3 bowel movements per week and/or at least one of the following constipation problems (straining during bowel movements, hard stools, feeling of incomplete emptying, gas/bloating, pressure/feeling of needing to defecate in the rectum).

Exclusion Criteria:

* Individuals with peripheral neuropathy,
* impaired foot skin integrity,
* flat feet or any foot deformity,
* and those using complementary treatments such as abdominal massage, acupressure, or acupuncture to relieve constipation were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Constipation Severity Scale | First week
  The Large Bowel Syndrome (LBS) consists of 16 questions in total and was developed to determine the frequency, intensity, and difficulty during defecation. The LBS comprises three sub-dimensions: "large bowel sluggishness," "fecal obstruction," and "pain." The highest possible score on the scale is 73. Scores for fecal obstruction range from 0-28, for large bowel sluggishness from 0-29, and for pain from 0-16.
Constipation Severity Scale | second week
  The Large Bowel Syndrome (LBS) consists of 16 questions in total and was developed to determine the frequency, intensity, and difficulty during defecation. The LBS comprises three sub-dimensions: "large bowel sluggishness," "fecal obstruction," and "pain." The highest possible score on the scale is 73. Scores for fecal obstruction range from 0-28, for large bowel sluggishness from 0-29, and for pain from 0-16.
Constipation Severity Scale | third week
  The Large Bowel Syndrome (LBS) consists of 16 questions in total and was developed to determine the frequency, intensity, and difficulty during defecation. The LBS comprises three sub-dimensions: "large bowel sluggishness," "fecal obstruction," and "pain." The highest possible score on the scale is 73. Scores for fecal obstruction range from 0-28, for large bowel sluggishness from 0-29, and for pain from 0-16.
Constipation Severity Scale | fifth week
  The Large Bowel Syndrome (LBS) consists of 16 questions in total and was developed to determine the frequency, intensity, and difficulty during defecation. The LBS comprises three sub-dimensions: "large bowel sluggishness," "fecal obstruction," and "pain." The highest possible score on the scale is 73. Scores for fecal obstruction range from 0-28, for large bowel sluggishness from 0-29, and for pain from 0-16.
Constipation Assessment Scale | Baseline
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | third day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | sixth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | ninth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | twelfth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | fifteenth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | eighteenth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | twenty-first day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | twenty-fourth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | twenty-seventh day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Constipation Assessment Scale | thirtieth day
  This is a scale consisting of 8 items in total, which inquires about abdominal bloating, gas, bowel sounds, fecal incontinence, feeling of fullness/pressure in the rectum, pain during defecation, small or lumpy stools, and the presence of an urgent need to defecate but inability to do so.
Overall Comfort Scale | Baseline
  It is a scale developed to assess an individual's need for comfort. In the evaluation of the scale, negatively worded items are reverse-coded and summed together with the positively worded items. The highest possible total score on the scale is 192, while the lowest possible total score is 48. The total score obtained is divided by the number of items on the scale to calculate the mean score, which is expressed on a scale ranging from 1 to 4. A score of 1 indicates low comfort, whereas a score of 4 indicates high comfort.
Overall Comfort Scale | thirty-fifth day
  It is a scale developed to assess an individual's need for comfort. In the evaluation of the scale, negatively worded items are reverse-coded and summed together with the positively worded items. The highest possible total score on the scale is 192, while the lowest possible total score is 48. The total score obtained is divided by the number of items on the scale to calculate the mean score, which is expressed on a scale ranging from 1 to 4. A score of 1 indicates low comfort, whereas a score of 4 indicates high comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patients have not given permission to share their data in this area.

REFERENCES:
- [Background] References Akyüz Özdemir, F., Can, G. 2024. "The Effect of Reflexology Socks in the Management of Opioid-Induced Constipation: A Randomized Controlled Trial", Cancer Nursing, 10-1097. Anjoman, A. Z., Mirghafourvand, M., Hughes, C., Havizari, S. 2021. "Effect of Foot Reflexology on Constipation: A Systematic Review and Meta-Analysis", [Dergi adı belirtilmemiş]. Arıkan Dirimen, G. 2016. "Palyatif Bakım Tanımı ve Felsefesi", Klinik Tıp Aile Hekimliği, 8(3), 1-5. Ayık Bıçak, D., Can, G. 2020. "Palyatif Bakım Hastalarında Konstipasyonun Yönetimi ve Akupresürün Etkinliği", Sağlık Akademisyenleri Dergisi, 7(2), 141-148. Barichella, M. et al. 2016. "Probiotics and Prebiotic Fiber for Constipation Associated with Parkinson Disease", Neurology, 87(12), 1274-1280. Bassotti, G., Battaglia, E. 2023. "Considerations for laxatives in terms of their interactions with other drugs", Expert Opinion on Drug Metabolism & Toxicology, 19(3), 121-123. Bayan, K. 2017. "Konstipasyona Güncel Yaklaşım", Klinik Tıp Bilimleri Dergisi, 5(2). Bharucha, A. E., Lacy, B. E. 2020. "Mechanisms, Evaluation, and Management of Chronic Constipation", Gastroenterology, 158(5), 1232-1249.e3. Camilleri, M. et al. 2017. "Chronic Constipation", Nature Reviews Disease Primers, 3, 1-19. Canbulat Şahiner, N., Demirgoz Bal, M. 2017. "A Randomized Controlled Trial Examining the Effects of Reflexology on Children With Functional Constipation", Gastroenterology Nursing, 40(5), 393-400. Candy, B. et al. 2015. "Laxatives for the Management of Constipation in People Receiving Palliative Care", Cochrane Database of Systematic Reviews, 5. Cevik, K. 2013. "Complementary and Alternative Therapy in Nursing: Reflexology", Ege Hemşirelik Fakültesi Dergisi, 29(2), 71-82. Cevik, K., Zaybak, A. 2018. "The Effect of Reflexology on Constipation in the Elderly", International Journal of Caring Science, 11(1), 309-318. Clark, K., Currow, D. C. 2013. "Constipation in Palliative Care: What Do We Use as Definitions and Outco